CLINICAL TRIAL: NCT03208049
Title: Predictors of Response to Insomnia Treatments for Gulf War Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDR 15-196; 1I01HX001839-01A2 (NIH)
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
Keywords: Insomnia; Behavioral Therapy; Cognitive Therapy; Sleep; Gulf War Veterans
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The investigators' hypotheses will be tested in a randomized parallel groups design. Randomization will be based on type of treatment assignment: either to Behavioral Therapy (BT) or to Cognitive Therapy (CT). After screening and randomization in the 2-week baseline phase, subjects will receive BT or CT in the 6-week treatment phase. There will be no more treatment after this point. At the end of the 6-week treatment, subjects will return to repeat the tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Therapy (BT) (Experimental): Behavioral Therapy (BT). The subject is prescribed a time in bed. After one week, depending on subject's daily sleep logs and adherence to treatment, the therapist suggests a new time in bed prescription. Napping is neither prescribed nor proscribed. However, if subjects find themselves having difficulty staying awake during the day, they are advised to take a brief (15 to 30 minutes) nap to ensure their safety. Subjects in BT are also provided with information about relevant elements of the science of sleep and healthy sleep practices.
  Interventions: Behavioral: Behavioral Therapy (BT)
- Cognitive Therapy (CT) (Experimental): Cognitive Therapy (CT). The CT treatment module is designed to meet three general goals: 1) identify dysfunctional sleep cognitions, 2) challenge their validity, and 3) replace them with more adaptive substitutes. Several specific techniques designed to meet these goals are discussed in materials distributed to subjects. Similar to BT, subjects in CT are provided with information about relevant elements of the science of sleep and healthy sleep practices.
  Interventions: Behavioral: Cognitive Therapy (CT)

INTERVENTIONS:
Behavioral: Behavioral Therapy (BT) — Behavioral Therapy will regulate time spent in bed based on information collected from sleep diaries during evaluation and treatment. Behavioral therapy is designed to improve sleep quality by matching opportunity for sleep to the amount of average total sleep calculated from sleep diaries. Once the quality of sleep has improved, sleep quantity is gradually increased by slowly increasing sleep opportunity. Stimulus control will strengthen the bed/sleep association by eliminating non-sleep activities from the bedroom.
  Arms: Behavioral Therapy (BT)
Behavioral: Cognitive Therapy (CT) — Cognitive Therapy is designed to identify maladaptive beliefs about sleep, challenge their validity, and replace them with more adaptive thinking patterns. This therapy aims to reduce sleep-related worry, anxiety, and fear. The treatment phase of the study lasts six weeks. During treatment, you will meet with a study therapist for a total of six sessions: once per week for six consecutive weeks. Each session lasts approximately 60 minutes.
  Arms: Cognitive Therapy (CT)

SUMMARY:
The purpose of this study is to evaluate the efficacy and effectiveness of Behavioral Therapy (BT) and Cognitive Therapy (CT) in Gulf War Veterans with insomnia. The Primary Outcome measure is the Insomnia Severity Index (ISI).

DETAILED DESCRIPTION:
The investigators' hypotheses will be tested in a randomized parallel groups design. Randomization will be based on type of treatment assignment: either to BT or CT. After screening and randomization in the 2-week baseline phase, subjects will receive BT or CT in the 8-week treatment phase. There will be no more treatment after this point.

All subjects will receive education about basic sleep hygiene as well as information about the science of sleep including sleep stages and sleep regulation.

Behavioral Therapy (BT). The subject is prescribed a time in bed. After one week, depending on subject's daily sleep logs and adherence to treatment, the therapist suggests a new time in bed prescription. Napping is neither prescribed nor proscribed. However, if subjects find themselves having difficulty staying awake during the day, they are advised to take a brief (15 to 30 minutes) nap to ensure their safety. Subjects in BT are also provided with information about relevant elements of the science of sleep and healthy sleep practices.

Cognitive Therapy (CT). CT is designed to meet three general goals: 1) identify dysfunctional sleep cognitions, 2) challenge the validity of these thoughts, and 3) replace them with more adaptive substitutes. Several specific techniques designed to meet these goals are discussed in materials distributed to subjects.

The investigators will continue to monitor progress post-treatment during the follow-up period. The complete package of outcome measures will be repeated at the follow-up session. The investigators will tell subjects the expected benefits of treatment is to continue and/or improve with time and the investigators will also encourage subjects to continue practicing the treatment instructions to maintain their progress after active treatment ends.

Subjects will be screened for eligibility via a phone interview and an in-person evaluation.

At the in-person evaluation, informed consent will be received and documented. The evaluation will consist of measures of cognitive impairment and depression, sleep disturbance, and medical and psychiatric history.

The following measures will be completed at weeks 1, 8, and 32: Insomnia Severity Index (ISI), Beck Depression Inventory (BDI); Beck Anxiety Inventory (BAI), 36-Item Short-Form Health Survey (SF-36), Functional Outcomes of Sleep Questionnaire (FOSQ), Multidimensional Fatigue Inventory (MFI), and Wake After Sleep Onset (WASO).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Gulf War Veterans of any racial or ethnic group
* Independent Living (not in nursing home or VA Extended Care facility)
* Subjective complaint of insomnia on the Insomnia Severity Index (ISI) greater than or equal to 10
* Subjects with PTSD will be included in this study as long as they do not meet criteria for depression described below
* Stable (3 weeks) CNS active medications that could significantly impact sleep or alertness
* Stable adult onset diabetes, controlled with insulin, oral medications or diet is acceptable
* Access to a device with video capabilities and ability to have the video on during study visits.

Exclusion Criteria:

Sleep-Related

* Excessive caffeine consumption (4 or more cups of coffee per day) and unable to reduce to 3 cups or less a day before lunch a day for 3 weeks prior to treatment
* Subjects will be initially screened by the Berlin Questionnaire (for sleep apnea)
* Those with responses suggestive of high risk for sleep apnea will be referred to Pulmonary Medicine for standard clinical screening including polysomnography
* Those where apnea is primarily responsible for their sleep complaints will be excluded
* Subjects working a rotating shift or an unconventional daytime shift (ending after 1830h) will be ineligible

Neuropsychiatric

* Hamilton Depression Scale (HDRS 24) and classified as high risk on the Columbia Suicide Severity Rating Scale (C-SSRS) in the past month
* Individuals are considered high risk if they have endorsement of either of the following on the C-SSRS:
* A positive endorsement, relative to the past 30 days, in the "Suicide Thoughts" section of item #4 (Have you had these thoughts and had some intention of acting on them) or item #5 (Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan?
* A positive endorsement, relative to the past 90 days, in the "Suicide Behavior" section of item #6 (Have you ever done anything, started to do anything, or prepared to do anything to end your life?)
* Current or lifetime history of a psychiatric disorder with primary psychotic features
* Current or lifetime bipolar disorder; prominent suicidal or homicidal ideation
* Current exposure to trauma, or exposure to trauma in the past 3 months
* Current or within the past 30 days: drug abuse or dependence (except nicotine)
* Current or expected cognitive behavior therapy for another condition (e.g.,: depression)
* Excessive alcohol consumption of >14 drinks per week or > 4 drinks per occasion
* Presence of any acute or unstable psychiatric condition(s) that requires referral for treatment
* Montreal Cognitive Assessment (MOCA) < 20 or Montreal Cognitive Assessment Blind (MOCA-Blind) < 15

Medical

* Acute or unstable chronic illness, including but not limited to:
* Uncontrolled thyroid disease
* Kidney disease
* Prostate or bladder conditions causing excessively frequent urination (> 3 times per night)
* Medically unstable congestive heart failure
* Angina
* Other severe cardiac illness as defined by treatment regimen changes in the prior 3 months
* Stroke with serious sequelae
* Cancer if < 1 year since end of treatment
* Asthma
* Emphysema
* Other severe respiratory diseases uncontrolled with medications
* Neurological disorders such as Alzheimer's disease, Parkinson's disease, and/or unstable epilepsy as defined by treatment regimen changes in the prior 3 months
* Unstable adult-onset diabetes will be excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A Yesavage, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tao Y, Peters ME, Drye LT, Devanand DP, Mintzer JE, Pollock BG, Porsteinsson AP, Rosenberg PB, Schneider LS, Shade DM, Weintraub D, Yesavage J, Lyketsos CG, Munro CA. Sex Differences in the Neuropsychiatric Symptoms of Patients With Alzheimer's Disease. Am J Alzheimers Dis Other Demen. 2018 Nov;33(7):450-457. doi: 10.1177/1533317518783278. Epub 2018 Jul 3. PMID 29969907
- [Result] Yesavage JA, Fairchild JK, Mi Z, Biswas K, Davis-Karim A, Phibbs CS, Forman SD, Thase M, Williams LM, Etkin A, O'Hara R, Georgette G, Beale T, Huang GD, Noda A, George MS; VA Cooperative Studies Program Study Team. Effect of Repetitive Transcranial Magnetic Stimulation on Treatment-Resistant Major Depression in US Veterans: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Sep 1;75(9):884-893. doi: 10.1001/jamapsychiatry.2018.1483. PMID 29955803
- [Result] McNerney MW, Sheng T, Nechvatal JM, Lee AG, Lyons DM, Soman S, Liao CP, O'Hara R, Hallmayer J, Taylor J, Ashford JW, Yesavage J, Adamson MM. Integration of neural and epigenetic contributions to posttraumatic stress symptoms: The role of hippocampal volume and glucocorticoid receptor gene methylation. PLoS One. 2018 Feb 7;13(2):e0192222. doi: 10.1371/journal.pone.0192222. eCollection 2018. PMID 29415058
- [Result] Hantke N, Adamson MM, Noda A, Lazzeroni LC, Beaudreau SA, Yutsis M, Fairchild JK, Kinoshita LM, Kong J, Sheng T, Waltzman D, Ashford JW, Yesavage JA. Posttraumatic Stress Disorder-Associated Cognitive Deficits on the Repeatable Battery for the Assessment of Neuropsychological Status in a Veteran Population. Fed Pract. 2021 Jan;38(1):28-34. doi: 10.12788/fp.0083. PMID 33574646

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Started | 26 | 24
Completed | 13 | 12
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT) | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.3) | 54.8 (6.0) | 56.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 21 | 19 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 25 | 21 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 12 | 7 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — Responses can range from zero to 4, where higher scores indicate more acute symptoms of insomnia; thus, the total score range is zero to 28.
  units on a scale | 17.0 (4.4) | 18.9 (3.7) | 17.9 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: Measure Description: This seven-item questionnaire asks respondents to rate the nature and symptoms of their sleep problems using a Likert scale. Questions relate to subjective qualities of sleep, including the severity of symptoms, the satisfaction with sleep patterns, the degree to which insomnia interferes with daily functioning, how noticeable the respondent feels his or her insomnia is to others, and the overall level of distress created by the sleep problem. Responses can range from zero to 4, where higher scores indicate more acute symptoms of insomnia; thus, the total score range is zero to 28.
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 26 | 24
score on a scale
  Week 1 | 17.0 (4.4) | 18.9 (3.7)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | 7.3 (4.9) | 10.9 (7.7)
  Week 32: number analyzed (Participants) | 13 | 12
  Week 32 | 7.9 (7.1) | 9.8 (6.4)

2. Secondary Outcome: Beck Depression Index (BDI)
Description: The Beck Depression Index (BDI) is a formative assessment and rating scale of depression. This self-report inventory, or 21-item questionnaire uses a Likert scale that measures the scale quality of magnitude of depression. Responses can range from zero to 3, where higher scores indicate more acute symptoms of depression; thus, the total score range is zero to 63.
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 25 | 23
units on a scale
  Week 1 | 11.2 (8.1) | 12.6 (9.4)
  Week 8: number analyzed (Participants) | 15 | 14
  Week 8 | 6.1 (8.3) | 10.4 (13.9)
  Week 32: number analyzed (Participants) | 11 | 10
  Week 32 | 7.7 (9.0) | 8.7 (7.5)

3. Secondary Outcome: Beck Anxiety Index (BAI)
Description: The Beck Anxiety Index (BAI) is a formative assessment and rating scale of anxiety. This self-report inventory, or 21-item questionnaire uses a Likert scale that measures the scale quality of magnitude of anxiety. Responses can range from zero to 3, where higher scores indicate more acute symptoms of depression; thus, the total score range is zero to 63.
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 26 | 24
units on a scale
  Week 1 | 10.2 (10.1) | 8.5 (8.0)
  Week 8: number analyzed (Participants) | 14 | 14
  Week 8 | 5.4 (6.6) | 7.6 (9.2)
  Week 32: number analyzed (Participants) | 12 | 12
  Week 32 | 7.8 (9.3) | 12.8 (13.4)

4. Secondary Outcome: SF 36-Item Health Survey 1.0 (SF-36)
Description: The 36-Item Short-Form Health Survey (SF-36) is a self-reported patient survey that measures health status and quality of life (QoL). It is used in a variety of settings, including clinical practice, research, and health policy evaluations. To score the SF-36, scales are standardized to obtain a score ranging from 0 to 100. Higher scores indicate better health status,
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 14 | 11
units on a scale
  Week 1 | 62.4 (18.8) | 62.1 (18.5)
  Week 8: number analyzed (Participants) | 9 | 6
  Week 8 | 71.4 (14.9) | 62.3 (23.9)
  Week 32: number analyzed (Participants) | 6 | 4
  Week 32 | 52.2 (15.9) | 56.5 (24.2)

5. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: The Functional Outcomes of Sleep Questionnaire (FOSQ) is a self-report tool that assesses how sleepiness affects a person's ability to perform daily activities. The score range is 5 to 20, with higher scores indicating better functioning.
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 25 | 22
units on a scale
  Week 1 | 15.3 (4.1) | 14.0 (3.3)
  Week 8: number analyzed (Participants) | 13 | 12
  Week 8 | 17.3 (3.7) | 14.8 (4.0)
  Week 32: number analyzed (Participants) | 10 | 9
  Week 32 | 16.9 (4.0) | 15.4 (4.4)

6. Secondary Outcome: Multidimensional Fatigue Inventory (MFI)
Description: The Multidimensional Fatigue Inventory (MFI), scores each item on a 5-point Likert scale. The total score for each of the five fatigue dimensions (general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue) is calculated by summing the relevant items, resulting in a range of 20 to 100, where a higher score signifies more severe fatigue.
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 25 | 22
units on a scale
  Week 1 | 61.8 (6.4) | 63.7 (4.9)
  Week 8: number analyzed (Participants) | 13 | 12
  Week 8 | 64.8 (8.4) | 64.8 (7.7)
  Week 32: number analyzed (Participants) | 9 | 8
  Week 32 | 64.6 (5.1) | 61.5 (6.6)

7. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: WASO refers to the total amount of time a person spends awake after initially falling asleep and before finally waking up in the morning, essentially measuring the duration of wakefulness periods that occur once sleep has begun; a high WASO indicates fragmented sleep and can be a sign of a sleep disorder like insomnia. WASO will be reported in minutes.
Time Frame: Week 1, Week 8, and Week 32
Population: Number analyzed decreased due to dropouts and missing data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
Number analyzed (Participants) | 19 | 23
Minutes
  Week 1 | 34.8 (47.8) | 41.5 (28.9)
  Week 8: number analyzed (Participants) | 10 | 12
  Week 8 | 6.5 (7.1) | 40.4 (20.8)
  Week 32: number analyzed (Participants) | 15 | 10
  Week 32 | 18.7 (9.6) | 8.5 (6.3)

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Behavioral Therapy (BT) | Cognitive Therapy (CT)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

LIMITATIONS AND CAVEATS:
The COVID pandemic limited subject recruitment and follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-08-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT03208049/Prot_000.pdf